CLINICAL TRIAL: NCT03760471
Title: A Collaborative Palliative and Oncology Care Intervention to Improve Symptoms and Coping During Treatment for Head and Neck Cancer
Brief Title: Palliative and Oncology Care Intervention: Symptom COACH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-1054
Record Dates: First submitted 2018-11-16; First posted 2018-11-30 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Cancer of Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Collaborative palliative and oncology care (Experimental)
  Interventions: Other: Evidenced-based symptom management and coping intervention

INTERVENTIONS:
Other: Evidenced-based symptom management and coping intervention — The intervention visits will focus on coping and the following symptoms prevalent during CRT: (1) pain and mucositis, (2) nausea, (3) constipation, (4) fatigue, (5) sleep disturbances, (6) xerostomia, (7) thick mucus, and (8) depression

SUMMARY:
The investigators propose to conduct the first pilot trial of a collaborative palliative and oncology care intervention for HNC patients receiving CRT to assess the feasibility and acceptability of the intervention. The intervention will incorporate weekly palliative care visits into standard oncology care targeting coping, mood, and symptom management.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients (≥18 years) with a diagnosis of HNC for which they are undergoing CRT
2. receiving all oncology care at Fox Chase Cancer Center (FCCC)
3. able to speak and read in English or with assistance from an interpreter

Exclusion Criteria:

1. patients with prior history of HNC for which they underwent CRT
2. patients with uncontrolled psychiatric disorders (psychotic disorder, bipolar disorder, major depression) or other co-morbid disease which the treating clinician believes prohibits informed consent or participation in the study
3. patients enrolled on other supportive care intervention trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who comply for acceptability of a collaborative palliative and oncology care intervention for patients with HNC receiving CRT | 12 months
  The intervention will be considered feasible if >50% of patients agree to enroll on the trial and if > 70% of the participants have at least half of the scheduled palliative care visits

SECONDARY OUTCOMES:
Percentage of patients with coping strategies longitudinally in relation to symptom burden, QOL, mood, and health care utilization | 11 weeks
  This exploratory aim will provide preliminary data on associations of coping with patient outcomes to power a larger trial. We will specifically examine whether approach-oriented coping is associated with lower symptom burden, higher QOL and mood, and reduced health care utilization (e.g fewer hospitalizations, fewer treatment breaks or reductions in chemotherapy dose intensity)

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No